CLINICAL TRIAL: NCT06028282
Title: Post-RAI Therapy Dosimetry and Quality Assessment of Target Tissue Dosing
Acronym: Varian
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SUNYUMU 1642552
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Thyroid Disease
Keywords: I-131
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Radioiodine I-131 (RAI): oral administration of radioiodine I-131 (RAI) to patients with well-differentiated thyroid cancer
  Interventions: Radiation: SPECT

INTERVENTIONS:
Radiation: SPECT — SPECT of thyroid traced with I-131

SUMMARY:
The goal of this clinical trial study is to(1) determine the tissue specific dose of I-131 taken up by residing thyroid issue in the thyroid bed post-RAI along with any other sites in the neck and mediastinum as well as (2) correlate the dose delivered to residual tissues in the neck with patient follow-up based clinical outcomes, biochemical and imaging data following RAI therapy in patients with well-differentiated thyroid cancer (DTC). The main question[s] it aims to answer are:

* [question 1] How can obtained whole body and planar images more adequately depict residual iodine-avid disease in the thyroid bed, neck or mediastinum?
* [question 2] How can we obtain information on the dose taken up by the tumor remnant to know how much radionuclide actually went to the residual disease/tissue? Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
In our current clinical practice, patients with well-differentiated thyroid cancer (DTC) who receive oral administration of radioiodine 1-131 (RAI) have whole body and planar images obtained 4-5 days post-treatment. These images often do not adequately depict residual iodine-avid disease in the thyroid bed, neck or mediastinum. Further, no information about what dose taken up by the tumor remnant is obtained and thus we are unable to know how much radionuclide actually went to the residual disease/tissue.

Using single photon emission computed tomography (SPECT)/CT we will be able to better localize and evaluate disease/tissue remnant or distant iodine-avid metastatic disease. In addition, using Varian Velocity Theranostics Dosimetry suite of software applications, we will be able to do dosimetry on post-RAI therapy patients and be able to better correlate clinical outcomes with tumor absorbed dose in addition to provide quality improvement for the radioiodine ablation.

ELIGIBILITY:
Inclusion Criteria:

* All minorities
* 18 years of age and older
* Ability to give consent
* Male or female
* Differentiated thyroid cancer (DTC)
* Previous total thyroidectomy
* Has either:

  * local lymph node metastases
  * distant mediastinal/cervical metastases
  * lung or osseous metastases as seen on prior imaging studies

Exclusion Criteria:

* Non-iodine avid disease
* Under 18 years of age
* Unable to give consent
* Pregnant women, Non-viable neonates or neonates of uncertain viability.
* Non-English-speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroid Disease
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-11-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Staging Accuracy and Improved Clinical Patient Care | 24 months
  In addition to providing a thorough evaluation for any iodine-avid disease in the thyroid bed, neck soft tissues and mediastinum, a SPECT/CT with a high-energy collimator will help better assess the clinical stage of disease at the time of RAI treatment. Thus, better staging accuracy will be obtained and this will improve clinical patient management

CONTACTS AND LOCATIONS:
Overall Officials: David Lubin, MD, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be the only information available for sharing purposes.

REFERENCES:
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Willowson KP, Eslick EM, Bailey DL. Individualised dosimetry and safety of SIRT for intrahepatic cholangiocarcinoma. EJNMMI Phys. 2021 Sep 14;8(1):65. doi: 10.1186/s40658-021-00406-2. PMID 34519900
- [Background] Lubin DJ, Tsetse C, Khorasani MS, Allahyari M, McGrath M. Clinical predictors of I-131 therapy failure in differentiated thyroid cancer by machine learning: A single-center experience. World J Nucl Med. 2021 Mar 15;20(3):253-259. doi: 10.4103/wjnm.WJNM_104_20. eCollection 2021 Jul-Sep. PMID 34703393
- [Background] Lassmann M, Reiners C, Luster M. Dosimetry and thyroid cancer: the individual dosage of radioiodine. Endocr Relat Cancer. 2010 Jun 3;17(3):R161-72. doi: 10.1677/ERC-10-0071. Print 2010 Sep. PMID 20448022
- [Background] Ferris HA, Williams G, Parker JA, Garber JR. Therapeutic implications of diffuse hepatic uptake following I-131 therapy for differentiated thyroid cancer. Endocr Pract. 2013 Mar-Apr;19(2):263-7. doi: 10.4158/EP12077.OR. PMID 23529347
- [Background] Alan Selcuk N, Toklu T, Beykan S, Karaaslan SI. Evaluation of the dosimetry approaches in ablation treatment of thyroid cancer. J Appl Clin Med Phys. 2018 Jul;19(4):134-140. doi: 10.1002/acm2.12350. Epub 2018 Jun 1. PMID 29858536
- [Background] de Koster EJ, Sulaiman T, Hamming JF, Schepers A, Snel M, van Velden FHP, de Geus-Oei LF, Vriens D. Radioiodine in Differentiated Thyroid Carcinoma: Do We Need Diagnostic Pre-Ablation Iodine-123 Scintigraphy to Optimize Treatment? Diagnostics (Basel). 2021 Mar 19;11(3):553. doi: 10.3390/diagnostics11030553. PMID 33808843